CLINICAL TRIAL: NCT07303114
Title: Missed Opportunities for HIV Screening in General Practice - A Retrospective Study
Brief Title: Missed Opportunities for HIV Screening in General Practice
Acronym: DepVIH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9478
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV infections; HIV Testing
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of new HIV diagnoses in France in 2022 is estimated to be between 4,200 and 5,700. Of these diagnoses, 43% of infections were detected at a late stage. The objective of this study is to identify missed opportunities for HIV testing in general practice and to understand the barriers to testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥18 years)
* diagnosed with HIV infection between January 1, 2021, and July 30, 2024

Exclusion Criteria:

-Subject who arrived in France in the year preceding or during the period between January 1, 2024, and July 30, 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years) diagnosed with HIV infection between January 1, 2021, and July 30, 2024
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of clinical signs suggestive of HIV infection | 1 year preceding HIV diagnosis
  This is a retrospective analysis of data on the presence or absence of clinical signs suggestive of HIV infection during the year preceding diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France